CLINICAL TRIAL: NCT06458556
Title: Transvaginal Radiofrequency Ablation With Morpheus Device for Treatment of Overactive Bladder.
Brief Title: Transvaginal Radiofrequency Ablation for Overactive Bladder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InMode MD Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DO613705A
Record Dates: First submitted 2024-06-04; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-05

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Non-blinded non-comparative pilot trial in which a total of 20 subjects with OAB are included. Subjects may include individuals with overactive balder and contraindications to alternative first- and second-line treatments, OAB and do not desire pursuing alternative first- and second-line treatments, refractory overactive balder, and urge predominate mixed urinary incontinence. Subjects will undergo treatment with the Morpheus system every 4 weeks for a total of 3 treatments. Follow up will occur at 3- month and 6-month intervals after the subjects first treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment with Morpheus (Experimental)
  Interventions: Device: Treatment with Morpheus

INTERVENTIONS:
Device: Treatment with Morpheus — Radiofrequency device treatment

SUMMARY:
To assess the effectiveness of transvaginal radiofrequency oblation by the Morpheus device at varying depths of penetration for improving urge predominate and urinary incontinence symptoms in women with overactive bladder .

ELIGIBILITY:
Inclusion Criteria:

* Age 18-85 years old
* Urinary incontinence for ≥ 3 months
* Reporting at least "moderate bother" on Item 2 on the Urinary Distress Inventor questioner, "Do you experience a strong feeling of urgency to empty your bladder" (on new patient paperwork)
* If mixed urinary incontinence, urge is reported predominant symptom on MESA score.
* >10 micturition per 24 hours and >3 urgency episodes on 3-ay bladder diary
* > 1 UUI episode on 3-day bladder diary
* Not currently taking anti-muscarinic or beta3 agonist therapy (after at least 2-week wash-out period)

Exclusion Criteria:

* Non-English speakers
* Severely impaired mobility or cognition
* Spinal cord injury or advanced/severe neurologic condition including Multiple Sclerosis, Parkinson's Disease
* Repair of pelvic organ prolapse in the previous 6 months
* Received intravesical botulinum injection within the previous 12 months
* History of implanted nerve stimulator for incontinence
* History of prior sling or vaginal mesh placement, UNLESS onset of UUI was completely unrelated to placement and severity was unaffected by mesh placement.
* Previous diagnosis of Interstitial cystitis
* Active pelvic organ malignancy
* History of pelvic radiation
* Urethral obstruction
* Urinary retention or prolonged catheter use
* Less than 12 months post-partum are currently pregnant, or plan to become pregnant in the following 12 months
* Untreated symptomatic urinary tract infection
* Unevaluated hematuria
* Medical instability
* Allergy to anesthetics used in the study
* Not available for follow-up in 6 months
* Participation in other research trials that could influence results of this study

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with overactive bladder
Enrollment: 17 (Actual)
Dates: Start 2023-06-19 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
To assess the effectiveness of radiofrequency (RF) ablation at varying depths of penetration for improving urge predominate urinary incontinence symptoms | 3 months
  Measured by The Urogenital Distress Inventory-6 (UDI-6). The Urogenital Distress Inventory-6 (UDI-6) assesses the severity of urogenital symptoms through six questions addressing frequent urination, urgency-related leakage, leakage during physical activity, small amounts of leakage, difficulty emptying the bladder, and pain or discomfort in the lower abdomen or genital region.
  0 = Not at all
  1. = Slightly
  2. = Moderately
  3. = Greatly The scores for each item are summed to give a total score, which ranges from 0 to 18. Higher scores indicate greater distress and symptom severity.
To assess the effectiveness of radiofrequency (RF) ablation at varying depths of penetration for improving urge predominate urinary incontinence symptoms | 3 months
  Measured by the Incontinence Impact Questionnaire Total Score. Normative values for a general population, 10% of whom scored above 4.8 on IIQ-7. Values obtained from patients with severe incontinence indicate that a score > 70 on the IIQ signifies a poor QOL. Lower scores on IIQ-7 may identify more females who are bothered by urinary incontinence. 7 items are divided into four domains (physical activity, travel, social relationships, emotional health). Item-level scores are rated on a four-point Likert scale (where 0=not at all and 3=greatly), determined by the self-reported impact of symptoms related to urinary incontinence.
  The average score of items responded to is calculated. The average, which ranges from 0 to 3, is multiplied by 33 1/3 to put scores on a scale of 0 to 100.

SECONDARY OUTCOMES:
To assess the effectiveness of RF ablation for improving subject-reported incontinence-related quality of life | 6 months
  Measured by The Urogenital Distress Inventory-6 (UDI-6). The Urogenital Distress Inventory-6 (UDI-6) assesses the severity of urogenital symptoms through six questions addressing frequent urination, urgency-related leakage, leakage during physical activity, small amounts of leakage, difficulty emptying the bladder, and pain or discomfort in the lower abdomen or genital region.
  0 = Not at all
  1. = Slightly
  2. = Moderately
  3. = Greatly The scores for each item are summed to give a total score, which ranges from 0 to 18. Higher scores indicate greater distress and symptom severity.
To assess the effectiveness of RF ablation for improving subject-reported incontinence-related quality of life | 6 months.
  Measured by the Incontinence Impact Questionnaire Total Score. Normative values for a general population, 10% of whom scored above 4.8 on IIQ-7. Values obtained from patients with severe incontinence indicate that a score > 70 on the IIQ signifies a poor QOL. Lower scores on IIQ-7 may identify more females who are bothered by urinary incontinence. 7 items are divided into four domains (physical activity, travel, social relationships, emotional health). Item-level scores are rated on a four-point Likert scale (where 0=not at all and 3=greatly), determined by the self-reported impact of symptoms related to urinary incontinence.
  The average score of items responded to is calculated. The average, which ranges from 0 to 3, is multiplied by 33 1/3 to put scores on a scale of 0 to 100.
To assess the effectiveness of RF ablation assess on urgency and associated life impact | 6 months
  Measured by the Medical, Epidemiologic, and Social Aspects of Aging (MESA ).The MESA questionnaire is consisted of 2 separate parts, with 6 questions concerning urgency urinary incontinence (UUI) and 9 concerning stress urinary incontinence (SUI).
  MESA SI (Stress Incontinence), theoretical scores ranged from 1 (mild) to 27 (severe).
  MESA UI (Urgency Incontinence), theoretical scores ranged from 1 (mild) to 18 (severe).
  Higher scores indicate more severe symptoms,

CONTACTS AND LOCATIONS:
Overall Officials: Mickey Karram, MD, Principal Investigator — Not affiliated
Locations (1):
- California Center for Pelvic Floor Disorders, Corona del Mar, California, United States

IPD SHARING:
Plan to Share IPD: No